CLINICAL TRIAL: NCT04831021
Title: Pre- or Per-dialytic Physical Exercise : a Cardioprotective Role?
Acronym: EXP DIAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: AIDER- Santé (Unknown); Avignon University (EA4278 - LaPEC) (Unknown); Pr Philippe OBERT (Unknown); Dr Claire MAUFRAIS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20_0462
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic kidney disease on dialysis; Physical exercise; Regional myocardial function; Myocardial stunning
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Myocardial Stunning | interventions — Dialysis; Exercise

STUDY DESIGN:
Intervention Model Description: All patients will be assigned to one dialysis session without physical exercise, one dialysis session with pre-dialytic physical exercise and one dialysis session with per-dialytic physical exercise in random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients issued from dialysis units (clinic) (Experimental)
  Interventions: Procedure: Dialysis without physical exercise; Procedure: Dialysis with pre-dialytic physical exercise; Procedure: Dialysis with per-dialytic physical exercise

INTERVENTIONS:
Procedure: Dialysis without physical exercise — Hemodialysis control condition
Procedure: Dialysis with pre-dialytic physical exercise — Patients will pedal for 30 minutes using a ergometer directly attached to the dialysis bed. The exercise will be performed 60 minutes before connection to hemodialysis.
Procedure: Dialysis with per-dialytic physical exercise — Patients will pedal for 30 minutes using a ergometer directly attached to the dialysis bed. The exercise will start 30 minutes after the start of dialysis.

SUMMARY:
This study aims at evaluating, in chronic kidney disease patients on dialysis, the effect of acute per- or pre-dialytic physical exercise on regional myocardial function and myocardial stunning, blood viscosity, arterial stiffness, variability of sinus rhythm, dialysis efficacy, inflammation, mineral and bone disorders, myokines and cardiac remodeling markers.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 20 to ≤ 79 years
* Undernourished patient according to the ARNOS score : ≥ 2
* No medical contraindication to physical activity
* Life expectancy greater than 6 months
* Patient on hemodialysis for more than 3 months
* Patients with relatively good echogenicity

Exclusion Criteria:

* Patient is participating in another Category I interventional study, or has participated in another interventional study within the past 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is under legal protection or under guardianship or curatorship
* It turns out to be impossible to give the patient informed information, or the patient refuses to sign the consent
* Pregnant, parturient or breastfeeding patient
* Patient with a contraindication to retraining
* Patient with valvular heart disease, arteriopathy of the lower limbs stage III and IV, amputation or knee or hip prosthesis
* Patient with musculoskeletal problems
* Patient with severe respiratory failure
* Paired sleep apnea syndrome
* BMI> 35
* Patient with automatic implantable defibrillator
* Heart transplant
* Uncontrolled high blood pressure
* Ejection fraction <45%
* Unstabilized coronaries
* Non-contributory stress ultrasound

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in regional myocardial function and myocardial stunning | Weekly over a period of 3 weeks

SECONDARY OUTCOMES:
Change in blood viscosity | Weekly over a period of 3 weeks
Change in arterial stiffness | Weekly over a period of 3 weeks
Change in sinus rhythm | Weekly over a period of 3 weeks
Change in dialysis efficacy | Weekly over a period of 3 weeks
Change in inflammatory markers | Weekly over a period of 3 weeks
Change in mineral and bone metabolism markers | Weekly over a period of 3 weeks
Change in myokines | Weekly over a period of 3 weeks
Change in cardiac remodeling markers | Weekly over a period of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul CRISTOL, MD, PhD, Principal Investigator — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE; François ROUBILLE, MD, PhD, Study Chair — CHU ADV, Department of Cardiology, Montpellier, FRANCE; Cécile TURC-BARON, MD, Study Chair — AIDER Santé, Montpellier, FRANCE; Jérôme ADDA, MD, Study Chair — CHU ADV, Department of Cardiology, Montpellier, FRANCE
Locations (2):
- France (2):
  - Lapeyronie Hospital clinical trials Department, Montpellier, Hérault
  - AIDER Santé, Montpellier

REFERENCES:
- [Derived] Josse M, Turc-Baron C, Patrier L, Connes P, Grandperrin A, Nottin S, Cristol JP, Hedon C, Roubille F, Maufrais C, Obert P. Acute Exercise before Dialysis Is as Cardioprotective as during Dialysis: A Randomized Controlled Trial. Clin J Am Soc Nephrol. 2025 Aug 12;20(9):1236-1246. doi: 10.2215/CJN.0000000767. PMID 40794519